CLINICAL TRIAL: NCT03744312
Title: Imaging Inflammation in Alzheimer's Disease With 11C-ER176
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Patrick Lao, Assistant Professor of Neurological Sciences, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR6570
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Inflammation; PET scans
MeSH Terms: conditions — Alzheimer Disease; Inflammation | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cognitive impairment (Experimental): Alzheimer's disease (mild cognitive impairment or mild stage Alzheimer's disease dementia)
  Interventions: Drug: 11C-ER176; Drug: Florbetaben
- No cognitive impairment (Active Comparator): Healthy Controls
  Interventions: Drug: 11C-ER176; Drug: Florbetaben

INTERVENTIONS:
Drug: 11C-ER176 — 11C-ER176 sticks to parts of the brain where there is inflammation. Past studies have shown that inflammation is present in the brains of patients with Alzheimer's disease. The purpose of this study is to determine if 11C-ER176 is able to accurately measure inflammation in patients with Alzheimer's disease.
  Other Names: [11C] ER176
Drug: Florbetaben — Florbetaben sticks to amyloid plaques, which are in the brain in Alzheimer's disease.
  Other Names: NeuraCeq

SUMMARY:
This study is being done to learn about inflammation in the brain of those with Alzheimer's disease (AD). The purpose of this study is to determine if 11C-ER176 is able to accurately measure inflammation in patients with Alzheimer's disease. Both patients (with either mild cognitive impairment (MCI) or Alzheimer's disease) and healthy controls (participants without memory complaints or impairment) will be included in this study.

DETAILED DESCRIPTION:
Inflammation likely plays a role in the damage to the brain caused by Alzheimer's disease.

Accurately measuring inflammation in the brain could provide new information about the mechanisms that cause Alzheimer's disease, and could help identify new treatments that reduce inflammation. Positron emission tomography (PET) imaging is a type of brain scanning method that allows investigators to measure small molecules in the brain. ER176-PET was recently developed as an improved method for measuring brain inflammation. However, ER176-PET has not yet been used in patients with Alzheimer's disease. The investigators propose to use ER176-PET imaging in subjects with mild cognitive impairment (a very early stage of Alzheimer's disease) or mild Alzheimer's disease to compare the amount of inflammation with that seen in older control subjects. The investigators will first use a "gold standard" method of measuring ER176 in brain that requires sampling arterial blood during the scan. The investigators will compare these results to those obtained using novel methods that don't require blood sampling. The investigators hope to show that ER176 is a useful tool for measuring inflammation in Alzheimer's disease, and that the investigators can develop a way to obtain ER176 PET scans that don't require arterial blood sampling.

This study uses a special type of scan called a PET scan to take pictures of the brain. During the PET scan, a special dye is injected into the body. Two types of dye will be used in this study: Florbetaben and 11C-ER176. Florbetaben sticks to amyloid plaques, which are in the brain in Alzheimer's disease. Florbetaben has been approved by the Food and Drug Administration to help diagnose Alzheimer's disease. 11C-ER176 sticks to parts of the brain where there is inflammation. Past studies have shown that inflammation is present in the brains of patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 and older
2. Meet criteria for either a) amnestic mild cognitive impairment or Alzheimer's disease, or b) have no cognitive impairment
3. If you are unable to provide informed consent, you must have a surrogate decision maker and be able to verbally assent to the study procedures
4. Written and oral fluency in English
5. Able to participate in all scheduled evaluations and to complete all required tests and procedures.
6. In the opinion of the investigator, you must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Past or present history of certain brain disorders other than MCI or AD.
2. Certain significant medical conditions, which make study procedures of the current study unsafe. Such serious medical conditions include uncontrolled epilepsy and multiple serious injuries.
3. Contraindication to MRI scanning
4. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
5. Exposure to research related radiation in the past year that, when combined with this study, would place you above the allowable limits.
6. Participation in the last year in a clinical trial for a disease modifying drug for AD.
7. Inability to have a catheter in your vein for the injection of radioligand.
8. Inability to have blood drawn from your veins.
9. Taking anticoagulant medication (e.g., warfarin).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lao, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon reasonable request from a qualified investigator.
Time Frame: Up to two weeks after review and approval of request.
Access Criteria: Investigator qualifications and previous work will be reviewed by PI. Subsequent email correspondence will relay technical criteria needed for access.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Impairment | No Cognitive Impairment
Started | 6 | 3
Completed | 6 | 1
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Screen fail | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data is analyzed for 7 out of the 9 enrolled participants. 2 participants either withdrew or screen failed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Impairment | No Cognitive Impairment | Total
Number analyzed (Participants) | 6 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 0 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: 11C-ER176 Total Distribution Volume
Description: Total distribution volume reflects the amount of TSPO (the inflammatory protein that 11C-ER176 sticks to) in the brain. This measure requires arterial blood sampling.
Time Frame: Up to one year from baseline
Population: Data is reflective of those with blood sampling only: 4 out of 6 cognitive impairment participants and 1 out of 1 no cognitive impairment participant. All 7 completers have 11C-ER176 imaging but only 5 have arterial blood sampling and therefore a Total Distribution Volume.
Measure: Mean (Full Range); unit: mL/cm^3
Arm/Group | Cognitive Impairment | No Cognitive Impairment
Number analyzed (Participants) | 4 | 1
mL/cm^3 | 6.27 [3.03 to 8.8] | 9.32 [9.32 to 9.32]

2. Secondary Outcome: 11C-ER176 Standardized Uptake Value Ratio
Description: The standardize uptake value ratio is the concentration of radioactivity measured from the 11C-ER176 positron emission tomography (PET) scan in the cortex compared to the uptake in the cerebellum (pseudo-reference region). This is a simplified quantification technique compared to the Total Distribution Volume, but is linearly related to it. Higher values indicate more neuroinflammation.
Time Frame: Up to one year from baseline
Population: Data is analyzed for completers only: 6 out of 6 cognitive impairment participants and 1 out of 1 no cognitive impairment participant. Completers here meaning they have 11C-ER176 imaging and SUVRs.
Measure: Mean (Full Range); unit: uptake value ratio
Arm/Group | Cognitive Impairment | No Cognitive Impairment
Number analyzed (Participants) | 6 | 1
uptake value ratio | 1.19 [1.10 to 1.38] | 1.22 [1.22 to 1.22]

ADVERSE EVENTS:
Time Frame: Up to one year.
Arm/Group | Cognitive Impairment | No Cognitive Impairment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 0/6 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03744312/Prot_SAP_000.pdf